CLINICAL TRIAL: NCT00367185
Title: Comparison of Melphalan-Prednisone(MP),MP-THALIDOMIDE,and Autologous Stem Cell Transplantation in the Treatment of Newly Diagnosed Elderly Patients With Multiple Myeloma.
Brief Title: Treatment of Newly Diagnosed Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFM 99-06
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2006-08-22 (Estimated); Status verified 2006-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Elderly patients; Thalidomide; Autologous transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
In multiple myeloma, combination chemotherapy with melphalan plus prednisone has been used since the 1960s and is regarded as the standard of care in elderly patients. We assess whether the addition of thalidomide to this combination or adapted high-dose chemotherapy, using a melphalan 100 mg/m2 -based regimen, would improve survival.

DETAILED DESCRIPTION:
Trial design This multicenter, randomized, controlled trial is conducted by the French Myeloma Intergroup(IFM) in elderly patients with previously untreated multiple myeloma. The primary objectives of the study are to compare the efficacy and safety of MP with MP-Thalidomide or with MEL100 (intermediate-dose melphalan 100 mg/m2 - based treatment). The secondary objective is to compare the efficacy of MP-Thalidomide vs MEL100.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III multiple myeloma according to Durie and Salmon criteria.
* Patients between 65 and 75 years of age
* Previously untreated patients

Exclusion Criteria:

* Prior history of another neoplasm (except basocellular cutaneous or cervical epithelioma)
* Primary or associated amyloidosis
* World Health organisation performance index of at least 3
* Significant renal insufficiency with creatinine serum levels of 5.0 mg per deciliter or more
* Cardiac or hepatic dysfunction
* Cerebral circulatory insufficiency
* Absolute contraindication to corticosteroids
* Peripheral neuropathy
* HIV or hepatitis B or C positivity
* Patients who had geographic, social or psychological conditions which might prevent adequate follow-up

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500
Dates: Start 2000-05; Study Completion 2005-10

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Best response rate
Progression-free survival
Survival after progression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves MARY, Study Director — U717 INSERM universite Paris7, Hopital Saint-Louis, Paris, France
Locations (1):
- Lille University Hospital, Lille, France

REFERENCES:
- [Derived] Facon T, Mary JY, Hulin C, Benboubker L, Attal M, Pegourie B, Renaud M, Harousseau JL, Guillerm G, Chaleteix C, Dib M, Voillat L, Maisonneuve H, Troncy J, Dorvaux V, Monconduit M, Martin C, Casassus P, Jaubert J, Jardel H, Doyen C, Kolb B, Anglaret B, Grosbois B, Yakoub-Agha I, Mathiot C, Avet-Loiseau H; Intergroupe Francophone du Myelome. Melphalan and prednisone plus thalidomide versus melphalan and prednisone alone or reduced-intensity autologous stem cell transplantation in elderly patients with multiple myeloma (IFM 99-06): a randomised trial. Lancet. 2007 Oct 6;370(9594):1209-18. doi: 10.1016/S0140-6736(07)61537-2. PMID 17920916